CLINICAL TRIAL: NCT04515316
Title: Development of A Room Temperature Atomic Magnetrode System for Telemetry of Epileptic Seizures
Brief Title: A Room Temperature Atomic Magnetrode System for Telemetry of Epileptic Seizures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-2363
Record Dates: First submitted 2020-04-06; First posted 2020-08-17 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy
Keywords: epilepsy; MEG
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Each feasibility group is of 20 persons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy adults (Experimental): Any adult, who is at least eighteen (18-70) years old.
  Interventions: Device: OPM sensors; Device: SQUID sensors
- Patients with intractable epilepsy (Experimental): Any clinical patient referred to us via the clinical MEG program, and who is at least eighteen (18-70) years old.
  Interventions: Device: OPM sensors; Device: SQUID sensors

INTERVENTIONS:
Device: OPM sensors — Optically-pumped magnetometers (OPM) sensors, which are based on optical probing of alkali atoms in the vapor phase at (or slightly above) room temperature, have recently demonstrated sensitivity levels comparable with SQUID magnetometers in the laboratory. These sensors require no cooling and can potentially be fabricated at much lower cost than SQUIDs. Beginning in the late 1990s, optically-pumped magnetometers began to be used for biomagnetic applications, first for measurement of heart magnetic fields and more recently for measurement of brain fields by several groups around the world.
Device: SQUID sensors — Magnetic sensors based on superconducting quantum interference devices (SQUIDs) have been the dominant sensor in the field of magnetoencephalography since its birth in the early 1970s. SQUIDs have exceptional sensitivity to enable the detection of these very weak signals. Current FDA-approved MEG devices contain liquid helium gas in a big container that is mounted over the head of the subject

SUMMARY:
This study is being done to help scientists learn about the use of a device called an atomic magnetometer. The device uses sensors called optically-pumped magnetometers (OPM) which function at room temperature. This research will compare the non-invasive brain imaging application of the OPM sensors to the present SQUID-based cryogenic sensor technique used in conventional Magnetoencephalography (MEG).

This study is being conducted in conjunction with the University of Colorado Boulder's Mechanical Engineering Department.

DETAILED DESCRIPTION:
Investigators at UC Boulder have an active program to develop "chip-scale" optically-pumped magnetometer (OPM) sensors, which combine high sensitivity with small size, low cost and low power operation. These sensors are an attractive alternative to superconducting quantum interference device (SQUID) magnetometers for the reasons outlined below, but remain largely unverified for use in biomagnetic applications. While considerable testing can be carried out without the use of humans, human testing is considered essential to encourage acceptance of this technology by the biomagnetic research community and more broadly by the medical community.

The goal of this research is to assess and validate how well the new types of sensors perform for non-invasive brain imaging and to optimize and improve their performance for imaging. The goal is to show that these sensors are not just more economical and easier to use, but also improve signal quality. In this project specifically, OPMs can prove usefulness for telemetry, which means that long-term measurements over several days are possible, in principle. This is important, since these non-invasive imaging with these OPM sensors might be able to use replace the invasive imaging with implanted electrodes (electrocoticography (EcoG) for pre-surgical mapping of epileptic seizures. The project proposes to compare the use of OPM and SQUID sensors during recording spontaneous and evoked brain activity in healthy human volunteers as well as in patients with intractable epilepsy. Two objectives: (1) to show that the patient can move with a confined area during measurements (this is currently not possible with rigid MEG systems) and (2) to show that images can be generated with a spatial resolution equivalent to that of internal electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Project A: Any adult subject, who is at least eighteen (18 - 70) years old.
* Project B: Any clinical patient referred to us via the clinical MEG program, and who is at least eighteen (18 - 70) years old.

Exclusion Criteria:

* ONLY applicable to Project A: have a history of neurological disorders (e.g., epilepsy, Parkinson disease, Alzheimer's disease, Autism, etc…).
* BOTH projects: have large amounts of metal or other magnetic field producing components present in their body or external to their body close to the measurement site, which are needed for normal functioning (e.g., metal implants, pacemakers, hearing aids, braces etc.). There is no harm to the subject with metal, it disturbs the sensor reading. Dental fillings are not excluded.
* BOTH projects: pregnant women.
* ONLY applicable to Project A: are not comfortable lying still for the time of the recording.
* BOTH projects: are unable to offer independent informed consent to study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evoked and Induced MEG with OPM and SQUID sensors in healthy controls | 1 day (during the brain scan)
  compare our own and published findings related to sensory-evoked brain activity using SQUIDs with results obtained with OPMs using the same paradigm and environment.
Spontaneous MEG with OPM and SQUID sensors in patients with epilepsy | 1 day (during the brain scan)
  compare the clinical findings related to the localization of interictal spike activity obtained during SQUID recordings as part of our clinical program with results from OPMs data collection on the same patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado School of Medicine - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No